CLINICAL TRIAL: NCT05105464
Title: A Multi-center, Open-label, Dose Escalation and Expansion, Phase I Study to Investigate the Safety, Tolerability, Pharmacokinetics (PK) Characteristic of SYHA1815 in Subjects With Unresectable Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study to Investigate the Safety of SYHA1815 in Subjects With Unresectable Locally Advanced or Metastatic Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Runshi Pharmaceutical Technology Co., Ltd (Industry)
Collaborators: Jilin Provincial Tumor Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SYHA1815-202001/PRO
Record Dates: First submitted 2021-09-13; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Locally Advanced Unresectable Carcinoma
Keywords: Locally advanced unresectable or metastatic solid tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Cohort (Experimental): Six dose levels will be tested. The dose-limiting toxicity (DLT) will be assessed from the first administration of SYHA1815 to the end of the first cycle (28 days).
  Interventions: Drug: SYHA1815
- cohort Expansion Cohort (Experimental): Once the expected effective dose is determined, four expansion cohorts will be started to further evaluate the safety, clinical activity and PK profile of SYHA1815.
  Interventions: Drug: SYHA1815

INTERVENTIONS:
Drug: SYHA1815 — Subjects will receive SYHA1815 orally.
  Other Names: SYHA1815 tablet

SUMMARY:
This is a multi-center, open-label, dose escalation and expansion, phase I study to investigate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) characteristics, preliminary efficacy of SYHA1815 in subjects with unresectable locally advanced or metastatic solid tumors. Once the expected effective dose is identified, the dose expansion study will be started to further evaluate the safety, clinical activity and PK profile of SYHA1815 in subjects with unresectable locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
This is a multi-center, open-label, dose escalation and expansion, phase I study to investigate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) characteristics, preliminary efficacy of SYHA1815 in subjects with unresectable locally advanced or metastatic solid tumors. The dose escalation study will include six dose cohorts starting at 2 mg/day. Once the expected effective dose is identified, the dose expansion study will be started to further evaluate the safety, clinical activity and PK profile of SYHA1815 in subjects with unresectable locally advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 to 75 years (inclusive)；
* Histologically or cytologically confirmed diagnosis of unresectable locally advanced or metastatic solid tumors (thyroid cancer, non-small cell lung cancer, gastric cancer [including gastroesophageal junction cancer], colorectal cancer, pancreatic cancer, soft tissue sarcoma, etc.), failure of standard treatment (disease progression or intolerance), or no alternative standard treatment or refusal of standard treatment;
* The subjects included in the dose expansion study should provide written biomarker test reports or tumor tissue samples to the central laboratory;
* The time interval between the last dose of anti-tumor drug and the first administration of SHYA1815 must meet the following conditions: ≥ 4 weeks for cytotoxic drugs, PD-1 / PD-L1, cellular immunotherapy; ≥2 weeks for oral molecular targeted drug therapy; ≥4 weeks for radiotherapy (≥ 2 weeks for palliative local radiotherapy for pain relief), and had recovered from the toxicities of radiotherapy; ≥2 weeks for anticancer Traditional Chinese medicine or Chinese patent medicine;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
* Life expectancy ≥ 12 weeks;
* At least one measurable lesion according to RECIST 1.1 at the screening phase;
* The organ function level and related laboratory values of the subjects must meet the following requirements within 7 days before the first dose of study drug (not receiving blood transfusion within 14 days before the first administration):

  1. Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L; Platelet count ≥ 75 × 10^9/L /L; Hemoglobin ≥ 90 g / L; the values of blood phosphorus and calcium are in normal range;
  2. Blood biochemistry: serum total bilirubin ≤ 1.5× upper limit of normal value (ULN); AST / ALT ≤ 3 ×ULN (≤ 5 ×ULN for liver metastasis); Serum creatinine ≤ 1.5 × ULN;
  3. Coagulation: Internationally standardized ratio (INR) or prothrombin time (PT) ≤ 1.5×ULN, activated partial thrombin time (APTT) ≤ 1.5×ULN;
* For women of childbearing potential: the serum pregnancy test within 7 days before the first administration must be negative, and female subjects are willing to take adequate contraceptive measures during the treatment period and for at least 3 months after the last dose of the study drug. Male subjects must agree to take contraceptive measures (non-drug or instrumental contraception) from the beginning of the study to at least 3 months after the last dose of study drug;
* Voluntarily participate in the study and sign the informed consent form.

Exclusion Criteria:

* The previous anti-tumor or surgical treatment history with any of the following conditions:

  1. Received the treatment of other intervention clinical studies with 4 weeks before the first dose of study drug;
  2. Had undergone major surgery within 4 weeks before the first dose of study drug or had not fully recovered from any previous invasive operation;
  3. Prior treatment of RET/FGFR inhibitors or small molecular kinase inhibitors with RET/FGFR as the main targets;
* Any unresolved toxicities from prior anti-tumor therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1, except for alopecia, pigmentation, previous chemotherapy-related neurotoxicity (≤ grade 2) and other adverse reactions judged no safety risk by the investigators;
* Subjects with symptomatic brain metastasis or meningeal metastasis, spinal cord compression or mental disorder, and asymptomatic brain metastasis can be enrolled (there is no disease progress within at least 4 weeks after radiotherapy and/or no neurological symptoms after surgical resection, and glucocorticoids, anticonvulsant drugs and mannitol are not required);
* Impaired cardiac function or clinically significant cardiovascular and cerebrovascular diseases, including any of the following:

  1. History of myocardial infarction, congestive heart failure (NYHA grade ≥ grade III), and unstable angina pectoris within 6 months prior to screening;
  2. Cerebrovascular disease occurred within 6 months before screening (except for transient ischemic attack (TIA), lacunar infarction with no clinical significance);
  3. Severe uncontrollable arrhythmia requiring medical treatment;
  4. Electrocardiogram (ECG) examination, female QTc interval>470 milliseconds (ms), male QTc interval>450 milliseconds (ms) according to Fridericia formula;
  5. The left ventricular ejection fraction is less than 50% according to cardiac ultrasound examination;
* History of active bleeding within 6 months before screening;
* Any serious or uncontrollable disease, and not suitable for this study as determined by the investigator;
* Any uncontrollable active infection that will prevent the subjects from receiving the study drug within 2 weeks prior to the first dose of study drug;
* HIV positive, HCV positive with HCV RNA quantity higher than the upper limit of normal value in the research center;
* Active hepatitis B infection, with the HBV DNA quantity higher than the upper limit of normal value of the research center;
* A history of any other malignant tumors within 5 years (except for effectively controlled non-melanoma skin basal cell carcinoma, cervical carcinoma in situ, and other malignant tumors that have been effectively controlled without treatment in the past 5 years;
* Subjects who have taken potent inhibitors and inducers of CYP3A4 liver metabolic enzymes within 2 weeks before the first administration and still need to continue to use such drugs;
* Women who are breastfeeding;
* Concomitant disease or condition that may interfere with the conduct of the trial, or that would pose an unacceptable risk to the subject in this trial in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2021-06-25 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose-limiting Toxicities | Baseline through 28 days after the first dose of study drug
  Number of participants with Dose-limiting Toxicities
Incidence of adverse events and SAEs | Up to 3 years
  Incidence of adverse events and SAEs defined by the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE V5.0).
Clinically significant changes from baseline in routine blood test | Up to 3 years
  Clinically significant changes from baseline in routine blood test
Clinically significant changes from baseline in blood biochemistry test | Up to 3 years
  Clinically significant changes from baseline in blood biochemistry test
Clinically significant changes from baseline in routine urine test | Up to 3 years
  Clinically significant changes from baseline in routine urine test
Clinically significant changes from baseline in coagulation function test | Up to 3 years
  Clinically significant changes from baseline in coagulation function test
Clinically significant changes from baseline in 12-lead electrocardiogram (ECG) | Up to 3 years
  Clinically significant changes from baseline in 12-lead electrocardiogram (ECG)
Clinically significant changes from baseline in vital signs examination | Up to 3 years
  Clinically significant changes from baseline in vital signs examination
Clinically significant changes from baseline in physical examination | Up to 3 years
  Clinically significant changes from baseline in physical examination

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 3 years
  Assessed by Blinded Independent Review Committee (IRC) per RECIST Version 1.1
Disease control rate (DCR) | Up to 3 years
  Disease control rate (DCR)
Duration of response (DOR) | Up to 3 years
  Duration of response (DOR)
Progression free survival (PFS) | Up to 3 years
  Progression free survival (PFS)
Time to maximum plasma concentration (Tmax) | Up to 3 years
  Time to maximum plasma concentration (Tmax)
Maximum Plasma Concentration (Cmax) | Up to 3 years
  Maximum Plasma Concentration (Cmax)
Plasma half-life (T1/2) | Up to 3 years
  Plasma half-life (T1/2)
Area under the plasma concentration-time curve from time 0 to time t (AUC0-t) | Up to 3 years
  Area under the plasma concentration-time curve from time 0 to time t (AUC0-t)
Area under the plasma concentration-time curve from time 0 to infinity (AUCinf) | Up to 3 years
  Area under the plasma concentration-time curve from time 0 to infinity (AUCinf)
Terminal disposition rate constant (λz) | Up to 3 years
  Terminal disposition rate constant (λz)
Apparent total clearance of the drug from plasma after oral administration (CL/F) | Up to 3 years
  Apparent total clearance of the drug from plasma after oral administration (CL/F)
Apparent volume of distribution during terminal phase after non-intravenous administration (Vz/F) | Up to 3 years
  Apparent volume of distribution during terminal phase after non-intravenous administration (Vz/F)
Change from baseline in serum phosphate | Up to 3 years
  Change from baseline in serum phosphate
Serum carcinoembryonic antigen (CEA) | Up to 3 years
  Serum carcinoembryonic antigen (CEA)
Calcitonin (thyroid cancer detection only) | Up to 3 years
  Calcitonin (thyroid cancer detection only)
Fibroblast growth factor 23 (FGF23) | Up to 3 years
  Fibroblast growth factor 23 (FGF23)
Vascular endothelial growth factor receptor 2 (sVEGFR2) | Up to 3 years
  Vascular endothelial growth factor receptor 2 (sVEGFR2)
Potential population who benefit from the study drug | Up to 3 years
  To evaluate the efficacy of the study drug in patients with different indications according to the results of anti-tumor response rate in the corresponding indications.
Correlation between the changes of RET/FGFR gene and efficacy | Up to 3 years
  The percentage of patients with RET/FGFR gene in patients who benefit from the study drug will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Huang Yanli, PD, Study Director — CSPC Zhongqi Pharmaceutical Technology (Shijiazhuang) Co., Ltd
Locations (1):
- Jilin Cancer Hospital, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No